CLINICAL TRIAL: NCT05285774
Title: Interest in the Implementation of a Systematic Protocol for the Dosage of the S100B Protein in the Reduction of the Use of Brain Scans for Patients With Mild Traumatic Brain Injury in the Emergency Room of Douai Hospital
Brief Title: Interest of the S100B Protein Assay in Mild Traumatic Brain Injuries at the DOUAI Hospital
Acronym: PS100BTCL
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Douai (Other)
Responsible Party: Sponsor
Other Study IDs: 01-2021-LJ3; IDRCB: 2021-A02163-38 (Other: ANSM)
Record Dates: First submitted 2022-02-25; First posted 2022-03-18 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Mild Brain Traumatic Injury; Compliance, Patient
Keywords: Protein S100B; Mild brain traumatic injury
MeSH Terms: conditions — Brain Concussion; Patient Compliance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective is to evaluate the feasibility and interest of setting up a protocol for the systematic measurement of the S100B protein in patients with mild traumatic brain injury admitted to the emergency room of Douai hospital in order to reduce the number of unnecessary brain scans. The main evaluation criterion is the percentage of patients admitted to the emergency department of Douai hospital for mild traumatic brain injury, whose protocol for the systematic measurement of the S100B protein would make it possible to avoid the realization of a brain scans for patients with a protein assay S100B ≤ 0.10 µg/L, carried out within 3h of the onset of MCT.

The systematic dosage of the S100B protein in the context of mild traumatic brain injury still does not appear in the recommendations for good practice in 2021. This study will contribute to the reflection on the use of the S100B protein in the development of new recommendations for good practice of mild traumatic brain injury support.

DETAILED DESCRIPTION:
This is an observational, prospective, monocentric study. This study concerns patients over 18 years of age treated in the emergency room of Douai hospital for mild traumatic brain injury treated within 3 hours following the head trauma according to the Jéle et al classification and who have no history of melanoma.

After verification of the patient's eligibility criteria for participation in this study, information relating to the research in order to obtain their authorization to participate in the research.

Once authorization has been obtained, an additional tube of blood is collected when drawing blood samples from the patient as part of their care.

Data are collected and a brain scan performed during the treatment and this is used to fill in the research data collection sheet.

The data used in this research come from the direct questioning of patients. They are recorded on a paper form or in a computerized medical record.

When the patient has been included in the trial the relevant data obtained from the direct questioning are taken from the sources indicated above and are entered on a data collection sheet specifically designed for this research.

The collection sheet will be placed in a dedicated tray and will be collected each week from the emergency room.The data will be compiled in EXCEL ® software secured by a password. This file is hosted on the Douai hospital center server with restricted access.

The files are protected by a password containing 8 characters (uppercase letters, lowercase letters and numbers), known only to the investigator, the person collecting the data, the clinical research assistant in charge of the study and the biostatistician in charge of data analysis.

To meet the main objective, the two-sided 95% confidence interval of the observed percentage of patients admitted to the emergency room of the Douai hospital for mild traumatic brain injury with a brain scan classified as avoidable by the S100B protein assay protocol will be calculated by the exact Clopper-Pearson method.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years having had a traumatic brain within 3h with Glasgow >13
* Patients having made a mild traumatic brain injury according to the Jehlé and Al classification:
* Either, amnesia of the facts > 30 minutes before the MCT (retrograde amnesia) or either, loss of consciousness or amnesia associated with one of the following mechanisms :
* Either pedestrian knocked down by a vehicle
* Either patients ejected from a vehicle
* Either fall from a height > 1 meter
* Either Age > 65 years old
* Either patients under anti platelet aggregation
* Patients informed about the study

Exclusion Criteria:

* Patients with a history of melanoma or in melanoma follow-up care
* Patients under guardianship or curatorship
* Patients deprived of liberty (prisoner)
* Patients not meeting MCT criteria
* Refusal to participate in the study
* Refusal to perform brain scan
* Glasgow Rating <13
* Unknown MCT Time
* Unclear patient history
* Polytraumatized
* Congenital or acquired coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study concerns patients aged over 18 years with no history of melanoma and treated in the emergency department of the CHD within 2h30 hours after a traumatic brain injury according to the Jehlé et al classification
Sampling Method: Probability Sample
Enrollment: 258 (Actual)
Dates: Start 2022-04-06 (Actual); Primary Completion 2023-08-06 (Actual); Study Completion 2023-08-06 (Actual)

PRIMARY OUTCOMES:
Measurement of the S100B protein to the emergency department of the Douai hospital | At 3 hours after MCT
  Percentage of patients admitted to the emergency department of the Douai hospital for MCT, whose protocol for the systematic measurement of the S100B protein would make it possible to avoid the realization of a brain scan for patients with a protein assay s100B ≤ 0.10 µg/L, carried out within 3h of the onset of MCT.

SECONDARY OUTCOMES:
Measurement of the S100B protein for a threshold ≤0.10 µg//l | At 3 hours after MCT
  Performance measures of the S100B protein for a threshold ≤0.10 µg//l: sensitivity, specificity, positive predictive value and negative predictive value.
Length of hospital stay | Immediatly after the procedure
  Evaluate the impact of adding this protocol to emergencies on the medical and paramedical team.

CONTACTS AND LOCATIONS:
Overall Officials: Justine HERENG, Principal Investigator — Centre Hospitalier de Douai
Locations (1):
- Centre Hospitalier de Douai, Douai, NORD, France

IPD SHARING:
Plan to Share IPD: No
There isn't a data sharing plan for this research

REFERENCES:
- [Background] Tiret L, Hausherr E, Thicoipe M, Garros B, Maurette P, Castel JP, Hatton F. The epidemiology of head trauma in Aquitaine (France), 1986: a community-based study of hospital admissions and deaths. Int J Epidemiol. 1990 Mar;19(1):133-40. doi: 10.1093/ije/19.1.133. PMID 2351508
- [Background] Mata-Mbemba D, Mugikura S, Nakagawa A, Murata T, Kato Y, Tatewaki Y, Takase K, Kushimoto S, Tominaga T, Takahashi S. Canadian CT head rule and New Orleans Criteria in mild traumatic brain injury: comparison at a tertiary referral hospital in Japan. Springerplus. 2016 Feb 25;5:176. doi: 10.1186/s40064-016-1781-9. eCollection 2016. PMID 27026873
- [Background] Bouvier D, Castellani C, Fournier M, Dauphin JB, Ughetto S, Breton M, Labbe A, Weinberg AM, Sapin V. Reference ranges for serum S100B protein during the first three years of life. Clin Biochem. 2011 Jul;44(10-11):927-9. doi: 10.1016/j.clinbiochem.2011.05.004. Epub 2011 May 13. PMID 21601568
- [Background] Unden J, Romner B. Can low serum levels of S100B predict normal CT findings after minor head injury in adults?: an evidence-based review and meta-analysis. J Head Trauma Rehabil. 2010 Jul-Aug;25(4):228-40. doi: 10.1097/HTR.0b013e3181e57e22. PMID 20611042